CLINICAL TRIAL: NCT06917482
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered BW-40202 in Healthy Subjects
Brief Title: A Study to Assess the Safety and Effects of the Investigational Drug BW-40202 in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Argo Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: BW-40202-1001
Record Dates: First submitted 2025-03-10; First posted 2025-04-08 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers Only
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm1: Single dose of BW-40202 (Active Comparator): 6 out of 8 participants randomized to cohort 1 will receive BW-40202
  Interventions: Drug: BW-40202 injection
- Arm2: Single dose of BW-40202 (Active Comparator): If deemed safe and tolerable by Safety Review Committee, dose level will escalate to cohort , 6 out of 8 participants within cohort 2 will be randomized to receive BW-40202
  Interventions: Drug: BW-40202 injection
- Arm3: Single dose of BW-40202 (Active Comparator): If deemed safe and tolerable by Safety Review Committee, dose level will escalate to cohort 3, 6 out of 8 participants within cohort 3 will be randomized to receive BW-40202
  Interventions: Drug: BW-40202 injection
- Arm4: Single dose of BW-40202 (Active Comparator): If deemed safe and tolerable by Safety Review Committee, dose level will escalate to cohort 4, 6 out of 8 participants within cohort 4 will be randomized to receive BW-40202
  Interventions: Drug: BW-40202 injection
- Arm5: Single dose of BW-40202 (Active Comparator): If deemed safe and tolerable by Safety Review Committee, dose level will escalate to cohort 5, 6 out of 8 participants within cohort 5 will be randomized to receive BW-40202
  Interventions: Drug: BW-40202 injection
- Arm 6: Placebo (Placebo Comparator): There will be 2 participants within each cohort be randomized to receive placebo.
  Interventions: Other: Sodium Chloride

INTERVENTIONS:
Drug: BW-40202 injection — BW-40202 is a conjugate drug, dosage form is solution for injection and route of administration is subcutaneous injection
  Arms: Arm1: Single dose of BW-40202; Arm2: Single dose of BW-40202; Arm3: Single dose of BW-40202; Arm4: Single dose of BW-40202; Arm5: Single dose of BW-40202
Other: Sodium Chloride — Placebo (sodium chloride injection) will be administered as Subcutaneous injection
  Arms: Arm 6: Placebo

SUMMARY:
This study will test the safety of a new drug called BW-40202 in healthy adults. The drug is a clear liquid given as an injection under the skin (subcutaneous injection). The study will test five different doses of BW-40202 compared to a placebo (saltwater solution).

Participants will be divided into five groups, with each group receiving a different dose of BW-40202 or placebo. In each group, eight people will be randomly assigned to receive either the drug (6 people) or placebo (2 people).

The Safety Review Committee will review the safety data before increasing the dose for the next group.

Study nurses or trained staff will give the injections. Pharmacy staff will keep records of how much drug each participant receives, any returned or destroyed doses, and any changes from the planned dosing schedule. These records will be securely stored and available for review.

ELIGIBILITY:
Key inclusion criteria:

1. Must have given written informed consent and be able to comply with all study requirements.
2. Males or females aged 18 to 60 years old, inclusive, at the time of informed consent.
3. BMI ≥18 and ≤32 kg/m2 with 50 kg <body weight ≤100 kg.

Key exclusion criteria:

1. Any clinically significant chronic medical condition or clinically significant abnormality in laboratory parameters that, in the opinion of the investigator, makes the subject unsuitable for participation in the study.
2. Hospitalization for any reason within 60 days prior to screening.
3. Any clinically significant acute condition such as fever (>38 degree centigrade) or acute respiratory illness within 14 days of study drug administration.
4. Systolic blood pressure (more than equal to) 140 mmHg and/or diastolic blood pressure (more than equal to) 90 mmHg after at least 5 minutes resting (seated or supine) at screening and Day -1(Repeat blood pressure measurement will be allowed at the discretion of the investigator).
5. Any liver function panel analyte value > 1.2 × upper limits of normal (ULN) which includes aspartate transaminase (AST), alanine transaminase (ALT), total bilirubin (TBIL), alkaline phosphatase (ALP) and gamma-glutamyl transferase (GGT) at screening.
6. International normalized ratio (INR) above 1.2 × ULN at screening or Day -1.
7. Single 12-lead electrocardiogram (ECG) with clinically significant abnormalities at screening or Day -1, asdetermined by the clinical investigator.
8. History or clinical evidence of alcohol abuse,
9. History or clinical evidence of drug abuse, within the 12 months before screening.
10. Donated or lost >200 mL of blood within 30 days prior to screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants experiencing at least one treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) from baseline to Day 169. To determine the incidenc of TEAEs and SAEs. | From first participant enrolled until Day 169 post-dose of last participant
  Incidence of TEAEs (%) = (number of subjects with TEAEs/Total number of subjects) *100 Incidence of SAEs (%) = (number of subjects with SAEs/total number of subjects)*100
Collecting the adverse events(AEs) up to D169 and the AEs will be categorized based on Medical Dictionary for Regulatory Activities (MedDRA) terms and clssified by System Organ Class (SOC) and Preferred Term (PT) for summary. | From first participant enrolled until Day 169 post-dose of last participant
  Adverse events (AEs) were coded using the latest MedDRA version available at the time of study commencement. All AEs were collected after drug administration and were considered TEAEs to be included in the summaries. Summary tables included the number of subjects (%) experiencing an event and the number of events. Subjects who experienced multiple AEs were only counted once in each category (system organ class [SOC] and preferred term [PT]), but all events were included in the event frequencies (categorical descriptive analysis).
  The TEAE summaries included:
  * Overall summary of TEAEs.
  * TEAE summary by SOC and PT.
  * TEAE summary of serious events by SOC and PT.
  * TEAE summary of study-drug related events by SOC and PT. TEAE summary by SOC, PT, and Toxicity Grading.
  * TEAE summary by SOC, PT, and relationship to study drug.
  * TEAE summary of events leading to study discontinuation by SOC and PT.
  * TEAE summary of Injection Site reactions.
Grading the TEAE and SAE based on severity and number of TEAEs and SAEs will be listed based on severity from baseline to Day 169. | From first participant enrolled until Day 169 post-dose of last participant
  Adverse events are graded based on severity:
  Mild (Grade 1): No significant impact on daily activities Moderate (Grade 2): Some interference with daily activities Severe (Grade 3): Significant impact on function Life-threatening (Grade 4): Immediate risk of death Fatal (Grade 5): Resulted in death.
  Severity distribution = (number of subjects with grade X TEAE/total TEAE cases) *100
Hematology results (concentration of Hemoglobin, g/L; Platelets, 10^9/L; Red blood cell count, 10^12/L) at each time point, including changes from baseline to Day 169 post dose will be summarized by treatment group. | From first participant enrolled until Day 169 post-dose of last participant
  The safety laboratory data will be summarized by visit and by treatment group, along with changes from baseline. The values that are below the lower limit or above the upper limit of the reference range will be flagged for safety. Those values or changes in values that are identified as being clinically significant will be flagged.
Coagulation results (Activated partial thermoplastic time, s; Prothrombin time, s) at each time point, including changes from baseline to Day 169 post dose will be summarized by treatment group. | From first participant enrolled until Day 169 post-dose of last participant
  The safety laboratory data will be summarized by visit and by treatment group, along with changes from baseline. The values that are below the lower limit or above the upper limit of the reference range will be flagged for safety. Those values or changes in values that are identified as being clinically significant will be flagged.
Chemistry results (concentration of Albumin, g/L; Alkaline Phosphatase, U/L; Alanine Amintransferase, U/L; Aspartate Aminotransferase, U/L;Direct Billirubin umol/L) at each time point from baseline to Day 169 will be summarized by treatment group. | From first participant enrolled until Day 169 post-dose of last participant
  The safety laboratory data will be summarized by visit and by treatment group, along with changes from baseline. The values that are below the lower limit or above the upper limit of the reference range will be flagged for safety. Those values or changes in values that are identified as being clinically significant will be flagged.
Urinalysis results（Epithelial cells, crystals, casts, bilirubin) at each time point, including change from baseline to Day 169 post dose will be summarized in the table by treatment group. | From first participant enrolled until Day 169 post-dose of last participant
  The safety laboratory data will be summarized by visit and by treatment group, along with changes from baseline. The values that are below the lower limit or above the upper limit of the reference range will be flagged for safety. Those values or changes in values that are identified as being clinically significant will be flagged.
Vital signs (blood pressures, millimeters of mercury) changes from Baseline values to Day 169 post dose will be summarized in the table by treatment group. | From first participant enrolled until Day 169 post-dose of last participant
  Abnormal physical examination findings will be listed.
Vital signs (heart rate, beats per minute) changes from Baseline values to Day 169 post dose will be summarized in the table by treatment group. | From first participant enrolled until Day 169 post-dose of last participant
  Abnormal physical examination findings will be listed.
Vital signs (temperature,degrees Celsius) changes from Baseline values to Day 169 post dose will be summarized in the table by treatment group. | From first participant enrolled until Day 169 post-dose of last participant
  Abnormal physical examination findings will be listed.
Changes in ECG (Mean heart rate, bpm; PR Interval,msec; QRS Duration, msec; QT interval, msec; RR interval, msec; QTcF Interval, msec; ) from Baseline to Day 169 post-dose will be summarized. | From first participant enrolled until Day 169 post-dose of last participant
  12-lead ECGs will be summarized by visit and by treatment group, along with the changes from baseline.The summary of overall interpretation findings table presented counts and percentages for the reported results at Baseline and Day 169/time point. Result categories were ordered as 'Normal', 'Abnormal Not Clinically Significant (NCS)' and 'Abnormal Clinically Significant (CS)' (categorical descriptive analysis).
By subject data listings will be created for all physical examination parameters(general appearance, head, neck, skin and others) from baseline to Day 169 post dose.. | From first participant enrolled until Day 169 post-dose of last participant
  Abnormal physical examination findings will be listed.
Vital signs (respiratory rate, times per minute) changes from Baseline values to Day 169 post dose will be summarized in the table by treatment group. | From first participant enrolled until Day 169 post-dose of last participant
  Abnormal physical examination findings will be listed.
Hematology results (White blood cell count and differential (absolute and % differential)) at each time point, including changes from baseline to Day 169 post dose will be summarized by treatment group. | From first participant enrolled until Day 169 post-dose of last participant
  The safety laboratory data will be summarized by visit and by treatment group, along with changes from baseline. The values that are below the lower limit or above the upper limit of the reference range will be flagged for safety. Those values or changes in values that are identified as being clinically significant will be flagged.
Coagulation results (International normalized ratio) at each time point, including changes from baseline to Day 169 post dose will be summarized by treatment group. | From first participant enrolled until Day 169 post-dose of last participant
  The safety laboratory data will be summarized by visit and by treatment group, along with changes from baseline. The values that are below the lower limit or above the upper limit of the reference range will be flagged for safety. Those values or changes in values that are identified as being clinically significant will be flagged.
Chemistry results (concentration of Calcium, mmol/L; creatine kinase, U/L; chloride, mmol/L; Gamma Glutamyl Transferase, U/L) at each time point from baseline to Day 169 will be summarized by treatment group. | From first participant enrolled until Day 169 post-dose of last participant
  The safety laboratory data will be summarized by visit and by treatment group, along with changes from baseline. The values that are below the lower limit or above the upper limit of the reference range will be flagged for safety. Those values or changes in values that are identified as being clinically significant will be flagged.

SECONDARY OUTCOMES:
maximum plasma concentration data (Cmax, ng/mL) of BW-40202 will be collected for all cohorts at the scheduled PK sampling timepoints. | From first patient enrolled until Day 8 post-dose of last patient.
  1. Collect Plasma Concentration Data Blood samples are collected at predetermined time points after drug administration.
     The drug concentration in plasma is measured at each time point.
  2. Plot the plasma concentration-time curve X-axis: time after drug administration y-axis: plasma drug concentration
  3. Identify the highest observed concentration locate the highest data point in the plasma concentration-time curve the corresponding drug concentration value is Cmax
Time to Maximum plasma concentration (Tmax, hr) of BW-40202 will be calculated (hr). T max(Time to Maximum Concentration) is the time at which the maximum observed plasma drug concentration ( Cmax) occurs after drug administration. | From first patient enrolled until Day 8 post-dose of last patient.
  1. Collect Plasma Concentration Data Blood samples are collected at predetermined time points after drug administration.
     The drug concentration in plasma is measured at each time point.
  2. Plot a Concentration-Time Curve The plasma drug concentration (C) is plotted on the Y-axis. Time post-dose (T) is plotted on the X-axis.
  3. Identify Cmax ⁡Determine the highest drug concentration observed in plasma. The corresponding time point is Tmax
Calculate the Area Under the Plasma Concentration-Time Curve (AUC, hr*ng/mL), to estimate the AUC beyond the last observed time point (AUC0-∞), the AUC from 0 to 24 hours and AUC from 0 to 48 hours. The AUC represents the total drug exposure over time. | From first patient enrolled until Day 8 post-dose of last patient.
  AUC (0-∞), Total drug exposure from time zero to infinity (extrapolated). The equation used to calculate Area Under the Plasma Concentration-Time Curve from Zero to Infinity AUC(0-∞) is based on the trapezoidal rule and extrapolation using the elimination rate constant (λz).
  AUC(0-24), Total drug exposure form time zero to 24 hours. The equation used to calculate Area Under the Plasma Concentration-Time Curve from Zero to 24 Hours (AUC₀-₂₄) is based on the trapezoidal rule and is called the Linear Trapezoidal Rule.
  AUC(0-48) , total drug exposure from time zero to 48 hours. The equation used to calculate Area Under the Plasma Concentration-Time Curve from Zero to 48 Hours AUC(0-48) is based on the trapezoidal rule and is called the Linear Trapezoidal Rule.
Calculate the time required for the plama concentration of a drug to decrease by 50% in the elimination phase. Which is called terminal elimination half-life (t1/2, hr) | From first patient enrolled until Day 8 post-dose of last patient
  1. Identify the Terminal Elimination Phase Plot a plasma concentration-time curve (log scale on Y-axis, linear scale on X-axis).
     Focus on the terminal elimination phase, where the concentration follows first-order kinetics (a straight line on a semi-log graph).
  2. Calculate the Elimination Rate Constant (Ke) Use the slope of the terminal phase of the log-transformed concentration-time curve
  3. Calculate the t1/2 using formula: t1/2=ln2/ke=0.693/ke.
Calculate the Urine output (Aet, mg), Aet (total amount of drug excreted in urine during each time interval) | From first participant being enrolled until 24 hours post-dose of last enrolled participant
  Total amount of drug excreted in urine from time t1 to t2 hours (for each urine time interval) Aet1 - t2=Cut1-t2*Vut-t2, where Vut1-t2 = the volume of urine collected from t1 to t2 and Cu t1-t2 = the concentration of drug in the collected urine. Parameters of interest are Ae0-4, Ae4-12, and Ae12-24.
Calculate the Urine output (Clr, L/h), the renal clearance measures the efficiency of drug elimination by the kidneys. | From first participant being enrolled until 24 hours post-dose of last enrolled participant
  Renal clearance calculated as CLr = CAe/Plasma AUC0-24. Ae=cumulative amount excreted in urine (mg). AUC0-24 = Area under the plasma concentration - timecurve from 0 to 24 hours (e.g. mg*h/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Zhuo Chang, MD. Ph.D, Study Director — Shanghai Argo Biopharmaceutical Co., Ltd.
Locations (2):
- Australia (2):
  - Q-Pharm Pty Ltd., Brisbane, Queensland
  - Nucleus Network Pty Ltd, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided